CLINICAL TRIAL: NCT00818636
Title: Expressive Writing for Co-Occurring Depression and Alcohol Misuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Carrie Dodrill, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R03AA016819-01A1 (NIH)
Record Dates: First submitted 2009-01-06; First posted 2009-01-08 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Depression; Alcohol, Drinking
Keywords: expressive writing; ruminating; ruminative thinking; experiential avoidance; depression; alcohol; drinking; emotional processing
MeSH Terms: conditions — Depression; Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Expressive Writing (Experimental): In addition to attending group therapy as usual, participants write about their feelings about an issue of their choosing three times during a two week period for at least 20 minutes each time.
  Interventions: Behavioral: Expressive writing (in addition to group therapy as usual).
- Treatment as Usual (Active Comparator): Participants attend group therapy as usual only.
  Interventions: Behavioral: Expressive writing (in addition to group therapy as usual).

INTERVENTIONS:
Behavioral: Expressive writing (in addition to group therapy as usual). — Participants in the expressive writing condition write about their feelings about an issue of their choosing three times, for at least 20 minutes each time, during a two week period.

SUMMARY:
***Please note that this study does not offer comprehensive treatment program for alcohol abuse or depression. Please do not contact the study staff if you are seeking psychological treatment. Further, this study is only enrolling people who are clients at Career and Recovery Resources, Inc., in Houston.

The hypothesis is that writing about feelings and thoughts will help people who are in group treatment feel less depressed and abuse alcohol less.

DETAILED DESCRIPTION:
Expressive writing applied to a variety of populations (e.g., HIV, cancer, PTSD, depression) has been associated with health improvements, reductions in symptoms of emotional distress, and one preliminary study found reductions in alcohol misuse among college students. Data suggest that expressive writing is a technique to facilitate emotional processing that can influence a number of clinical outcomes by facilitating cognitive restructuring (Hunt, 1998; Pennebaker, 2004). In addition to examining cognitive content change following expressive writing, we believe the effects of emotional writing on mood and drinking may involve two additional processes that have been found significant for both depression and alcohol misuse, namely experiential avoidance and ruminative thinking. We hypothesize that expressive writing will lead to less drinking and enhanced mood by reducing: (1) negative thought content, (2) experiential avoidance of unpleasant private events (e.g., negative thoughts, feelings, bodily sensations), and (3) ruminative thinking.

ELIGIBILITY:
***Please note that this study does not offer comprehensive treatment program for alcohol abuse or depression. Please do not contact the study staff if you are seeking psychological treatment. Further, this study is only enrolling people who are clients at Career and Recovery Resources, Inc., in Houston.

Inclusion Criteria:

* Enrolled in group therapy program at Career and Recovery Resources, Inc.
* Must be at least 18.
* Willing and able to participate in the study through the one month follow up.
* Able to provide the contact information of at least two people who can generally locate their whereabouts.
* Speak English fluently.

Exclusion Criteria:

* Inability to read, write, speak English.
* History of bipolar or psychotic disorders.
* Severe medical, cognitive and /or psychiatric impairment that precludes cooperation with study protocol.
* Substance withdrawal symptoms requiring medical attention.
* Currently receiving other individual psychosocial therapy outside of C&R for substance abuse or other psychiatric conditions with the exception of AA, NA or CA.
* Impending incarceration or other factor that would create inability or unwillingness to participate in the 6 week long study period (e.g., halfway house or other aftercare program restrictions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory, Second Edition | Baseline, Post-writing (2 weeks post-baseline), and One Month Follow-Up (Six weeks post-baseline)

SECONDARY OUTCOMES:
Number of Alcoholic Drinks Consumed | 30 days pre-baseline compared to 30 days post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Carrie L Dodrill, Ph.D., Principal Investigator — The University of Texas Health Science Center at Houston- ** This contact information should not be used for counseling or informational purposes**; Angela L Stotts, Ph.D., Study Chair — The University of Texas Health Science Center at Houston- ** This contact information should not be used for counseling or informational purposes**
Locations (1):
- Career and Recovery Resources, Inc., Houston, Texas, United States

REFERENCES:
- [Background] Frattaroli J. Experimental disclosure and its moderators: a meta-analysis. Psychol Bull. 2006 Nov;132(6):823-65. doi: 10.1037/0033-2909.132.6.823. PMID 17073523
- See also: Please note that this study does not offer comprehensive treatment program for alcohol abuse or depression. Please do not contact the study staff if you are seeking psychological treatment. This study is only enrolling people at Career and Recovery. — http://www.clinicaltrials.gov